CLINICAL TRIAL: NCT02113696
Title: The Effect of ω-3 Polyunsaturated Fatty Acids (Eicosapentaenoic Acid and Docosahexanoic Acid) on Morbidly Obese Patients
Brief Title: Intake of Omega 3 in Morbidly Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidade Católica do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: primary
Record Dates: First submitted 2014-03-27; First posted 2014-04-15 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Morbid Obesity
Keywords: morbid obesity; BMI at or above 4O kg/m2; ingestion of omega 3; inflammatory cytokines; biochemical factors; anthropometric factors
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo group (Experimental): Placebo Capsules
  Interventions: Dietary Supplement: Placebo Capsules
- Omega 3 intake (Experimental): Omega 3 intake, morbid obesity
  Interventions: Dietary Supplement: Omega 3 intake, morbid obesity

INTERVENTIONS:
Dietary Supplement: Omega 3 intake, morbid obesity — Individuals of both sexes with ages between 18 and 65 years took 3g of omega 3, and 1.8g eicosapentaenoic acid (EPA) and 1.2g docosahexanoic acid (DHA) for 8 weeks.
  Arms: Omega 3 intake
Dietary Supplement: Placebo Capsules — They received gelatin (colorless) capsules. A nutritional evaluation was performed, a 24-h recordatory was applied to verify macro and micronutrients intake, biochemical evaluation before and after the intervention. Macro and micronutrients were calculated using the Avanutri 2.0 system. Clinical history was verified through a questionnaire previously filled out by a physician.
  Arms: Placebo group

SUMMARY:
Ingestion of capsules of omega 3 EPA and DHA, with 1.8 g of EPA and 1.2 g DHA for morbidly obese patients, will improve the inflammatory status? C-reactive protein? Weight?

DETAILED DESCRIPTION:
Intake of EPA and DHA for the management of morbid obesity in capsules

- Reduction of inflammatory factors such as adipokines, glucose, C-reactive protein, cholesterol, weight, BMI. Will be 2 groups: cases and controls. The cases will intake of omega 3 capsules and placebo control.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18-65 years,
* BMI > 40 kg/m2 (or > 35 kg/m2 with comorbidities),
* ambulatory, receiving an oral diet,
* with a diagnosis of metabolic syndrome,
* and who signed a Term of Free and Informed Consent.

Exclusion Criteria:

* Systemic inflammatory response syndrome,
* coma or compromised organ,
* fever or infection foci,
* cancer with or without chemotherapy and radiotherapy,
* radiotherapy, inflammatory diseases of the gastrointestinal tract,
* transplant, trauma, surgery or hospital stay in the past 30 days
* use of steroids or non-steroid anti-inflammatory or immunomodulators agents or antibiotics,
* or those refusing to take part in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Decrease of inflammatory levels on blood | 08 weeks
  expected from this study verify inflammatory factors such as adipokines, glucose, c reactive protein, lipid profile, triglycerides, and anthropometric data as visceral fat, weight, BMI, in both groups, control and intervention, to see the action of the capsules of omega 3.patient may withdraw any time from ingestion of capsules, and the same will be provided by the laboratory Vitamed, which is regularized with the supervisory bodies and food security of Brazil

SECONDARY OUTCOMES:
Decrease of weight | 08 weeks
  The weight will be measured before and after the intake of omega 3.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio C Motin, orientador, Study Director — Centro de Obesidade Mórbida da Pontificia Universidade Católica do RS